CLINICAL TRIAL: NCT01176734
Title: The Treatment of Tinnitus With Transcutaneous Non-invasive Vagus Nerve stimulation-a Controlled Randomized Pilot Study Assessing Safety, Compatibility and Clinical Performance
Brief Title: The Treatment of Tinnitus With Transcutaneous Non-invasive Vagus Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: cerbomed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cMPsTIN01
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Tinnitus
Keywords: Pulsatile Tinnitus; Ringing-Buzzing-Tinnitus; Spontaneous Oto-Acoustic Emission Tinnitus; Tensor Palatini Induced Tinnitus; Tensor Tympani Induced Tinnitus; Tinnitus of Vascular Origin; Tinnitus, Clicking; Tinnitus, Leudet; Tinnitus, Leudet's; Tinnitus, Noise Induced; Tinnitus, Objective; Tinnitus, Spontaneous Oto-Acoustic Emission; Tinnitus, Subjective; Tinnitus, Tensor Palatini Induced; Tinnitus, Tensor Tympani Induced; Vascular Origin Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active t-VNS (Experimental): active t-VNS
  Interventions: Device: tVNS-Device

INTERVENTIONS:
Device: tVNS-Device — Active treatment with the t-VNS device.

SUMMARY:
The t-VNS STv3 device is a non-invasive, transcutaneous neurostimulator for influencing the afferent branches of the nervus vagus around the human ear. The clinical trial is designed as a a pilot study addressing the treatment of tinnitus with transcutaneous vagus nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tinnitus defined as a tinnitus over more than six months
* ≥31 points in the tinnitus questionnaire according to Goebel and Hiller
* Written informed consent
* Both gender, aged from 18 -75 years
* If the subject takes psychoactive medication (e.g antidepressants, anticonvulsives) therapy must be stable for at least 10 days. If a treatment with neuroleptics is necessary, only olanzapine and quetiapine should be used. The therapy should be constantly though a necessary change in medication is no reason for exclusion of the subject.

Exclusion Criteria:

* Objective tinnitus
* Participating in other tinnitus treatments within 3 months before study start
* Missing informed consent
* Pregnancy
* Bronchial asthma in medical history
* Clinically relevant internistic, neurological or psychiatric diseases
* Abuse of drugs or alcohol until 12 weeks before enrollment in the study
* Indications of structural impairment of the basal ganglia or the brain stem
* Active implants (e.g. cochlea implants, VNS, pacemaker)
* Constant all-day use of hearing instruments or noisers on the left the part-time use in special situations (e.g. watching TV is no exclusion criteria
* All dermatologic and infectious diseases which affect the area around the pinna and the ear canal
* Severe malformation of the pinna
* Other circumstances that in the opinion of the investigator might be an obstacle for enrolling the subject

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety, feasibility and effectiveness of t-VNS® stimulation | 24 weeks
  Determination of safety, feasibility and effectiveness of t-VNS measured by tinnitus score according to Goebel and Hiller between baseline and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Principal Investigator — University of Regensburg
Locations (1):
- Klinik für Psychiatrie und Psychotherapie Bezirksklinikum Regensburg Universitätsstr. 84 93053 Regensburg E-mail: Berthold.Langguth@medbo.de Tel.: 0941 941 2099 Fax.: 0941 941 2025 Dr. med Michael Landgrebe, Klinik für Psychiatrie und Psychotherapie Bezir, Regensburg, Bavaria, Germany

REFERENCES:
- [Derived] Kreuzer PM, Landgrebe M, Resch M, Husser O, Schecklmann M, Geisreiter F, Poeppl TB, Prasser SJ, Hajak G, Rupprecht R, Langguth B. Feasibility, safety and efficacy of transcutaneous vagus nerve stimulation in chronic tinnitus: an open pilot study. Brain Stimul. 2014 Sep-Oct;7(5):740-7. doi: 10.1016/j.brs.2014.05.003. Epub 2014 Jun 4. PMID 24996510